CLINICAL TRIAL: NCT00380614
Title: A Randomized Controlled Trial of Lamivudine in Acute Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maulana Azad Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ethical/Path/GBPH/805
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis B
Keywords: Acute Hepatitis B, Lamivudine
MeSH Terms: conditions — Hepatitis B | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine

SUMMARY:
Since a proportion of patients with Acute Viral Hepatitis-B develop severe hepatitis and fulminant hepatic failure, it is logical to believe that a rapid reduction in the HBV DNA levels by using antiviral agents could result in a less intense host response against the hepatitis B virus. However, the experience with lamivudine treatment of immunocompetent patients with AVH-B is limited.The aim of the present study was to evaluate the efficacy, utility and safety of lamivudine in treating immunocompetent patients with AVH-B.

DETAILED DESCRIPTION:
The diagnosis of acute hepatitis B was based on recent onset acute illness including prodromal symptoms, jaundice and other typical symptoms. The laboratory investigations supporting the diagnosis of acute hepatitis included the presence of >2.5 times the upper limit of serum alanine aminotransferase (ALT) and serum bilirubin, and positive IgM anti-HBc test. Ultrasound, and esophagogastroduodenoscopy was done to look for any evidence of chronic liver disease. All patients had normal alpha-fetoprotein levels.

Co-infection with hepatitis A, C, D, E and human immunodeficiency virus (HIV) infection was looked for by appropriate serologic tests conducted within 7 days of presentation.

Patients with co-infection, a history of hepatotoxic drug intake or alcohol use >20g/day, or any evidence of chronic liver disease in the past, at presentation or during follow-up were excluded. Patients were also excluded if they had serum bilirubin < 5 mg/dl at presentation.

Patients were classified as severe AVH-B if they fulfilled any two of the following criteria: (1) hepatic encephalopathy; (2) serum bilirubin ≥10.0 mg/dl; and (3) international normalized ratio (INR) ≥1.6.

The patients were randomized into 2 groups: Group 1: Treatment with lamivudine 100 mg daily for 3 months, Group 2: Placebo. Randomization was done using random number table. The initial study and randomization was planned to enroll 120 patients or continue the study till three years, whichever was earlier. Individual rather than block randomization was done The investigators as well as the patients were blinded to the randomisation. The patients in the placebo group received a placebo pill.

All patients were monitored during treatment for clinical evidence and grade of hepatic encephalopathy, impaired coagulation (abnormal international normalized ratio, IINR), AST/ALT, serum albumin bilirubin levels every week for the first month and then monthly. HBV serology, including serum HBsAg, HBeAg, and anti-HBe were checked at baseline and every 3 months. Anti-HBs titres were checked at 6 and 12 months. Quantitative HBV DNA assay was performed on day 0, day 4, week 1, week 2, week 3, week 4, then every month for the next 2 months and then every 3 months for 12 months.

All patients were followed for at least 12 months after the onset of AVH-B. Development of protective anti-HBs(>10 IU/L) was specifically looked for.

Exacerbation of chronic hepatitis B was excluded by investigating thoroughly for any evidence of chronic liver disease by Ultrasound, Upper GI endoscopy, or low albumin at presentation. Ultrasound was repeated at 6 and 12 months, and if there was any suspicion Upper GI endoscopy was also repeated. LFTS were done at every hospital visit.

HBsAg, HBeAg, IgM anti-HBc, anti-HBs, and anti-HBe were tested by commercially available enzyme-linked immunoassays. Serum quantitative HBV DNA assay was performed by use of an ultra sensitive Hybrid capture assay [Digene Labs, USA] that has a lower limit of detection of 4,700 copies/ml. An arbitrary value of 4,700 copies/ml was assigned to values < 4,700 copies/ml for analysis purposes. In such patients HBV DNA was done by an in-house qualitative PCR test to indicate negativity or positivity of viral DNA. The lower limit of detection was 600 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute hepatitis B
* Bilirubin > 5 mg/dl at presentation.

Exclusion Criteria:

* Patients with co-infection, a history of hepatotoxic drug intake or alcohol use >20g/day, or any evidence of chronic liver disease in the past, at presentation or during follow-up

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-01; Study Completion 2005-03

PRIMARY OUTCOMES:
clinical improvement
biochemical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G.B. Pant Hospital, New Delhi, India
Locations (1):
- G.B. Pant Hospital, New Delhi, National Capital Territory of Delhi, India